CLINICAL TRIAL: NCT06884163
Title: Characterization of the Immune Signature of Chronic Hand Eczema With an Innovative Approach Combining Spatial Transcriptomics and Single Cell Spatial Proteomics
Brief Title: Immune Signature of Chronic Hand Eczema Unveiled by Spatial Transcriptomics and Single-Cell Proteomics
Acronym: ECMANDO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7219
Record Dates: First submitted 2025-03-03; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Hand Eczema
Keywords: atopic; biopsy; itch
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Masking Description: comphrensive spatial transcriptomic on skin biopsies of chronic hand eczema aims to describe differerent immune endotypes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients affected by chronic hand eczema (Other): Patients with a diagnosis of chronic hand eczema
  Interventions: Genetic: comprhensive spatial transcriptomic profile on lesional skin biopsies

INTERVENTIONS:
Genetic: comprhensive spatial transcriptomic profile on lesional skin biopsies — Spatial transcriptomics (Visium, 10X Genomics) will be used to analyze gene expression of chronic eczema derived from lesional skin biopsies

SUMMARY:
The study explores the immune landscape of chronic hand eczema using spatial transcriptomics and single-cell proteomics, offering new insights into disease mechanisms and potential therapeutic targets.

DETAILED DESCRIPTION:
Patients aged 18 to 65 affected with chronic hand eczema will be included in the study. As clinical practice, severity of chronic hand eczema will be evaluated by validated scores as HECSI, DLQI, and NRS itch. Moreover patch tests will be performed. Skin biopsies will also be performed to confirm the diagnosis.

This study utilizes spatial transcriptomics and single-cell spatial proteomics to analyze biopsies of chronic hand eczema. It aims to identify distinct inflammatory cell subgroups and molecular markers that define the immune landscape of chronic hand eczema.

By comparing endogenous (atopic dermatitis, dyshidrotic eczema, idiopathic forms) and exogenous (allergic/irritant) chronic hand eczema, the research wants to describe specific immune endotypes and potential therapeutic targets.

The study also includes idiopathic chronic hand eczema subtypes, such as pompholyx and hyperkeratotic eczema, to clarify immune profiling and improve treatment strategies. By identifying molecular signatures unique to each chronic hand eczema subtype, this research could lead to more personalized and effective therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected with chronic hand eczema of endogenous and/or exogenous origin, age from 18 to 65 years
* Patients affected with eczema located on the hands for at least 3 months or with ≥ 2 disease flare-ups in the last year.
* Patients affected with atopic dermatitis affecting the hands and other areas of the body, provided the eczema lesions involve less than 30% of the body surface area.

Exclusion Criteria:

* Concurrent or previous treatment with immunosuppressants, except for short courses of systemic corticosteroids (less than one month of continuous treatment), or biologic agents that may affect the clinical aspects or progression of chronic hand eczema.
* Patients who have received systemic corticosteroids within one month prior to enrollment in the study.
* Patients using topical corticosteroids or calcineurin inhibitors within one week of study enrollment (this time frame is considered to provide a good balance between potential residual pharmacological effects and ethical considerations).
* Patients with chronic hand eczema of mixed etiology (e.g., allergic and atopic) or those considered "etiologically unclassifiable" will not be included in the data analysis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
spatial proteomics analysis | through study completion, an average of 2 years
  Based on the gene expression profile obtained from the spatial transcriptomics analysis (Visium 10X Genomics), a subset of markers of interest will be selected. These markers will then be analyzed using spatial proteomics on the same lesional sections of chronic hand eczema

CONTACTS AND LOCATIONS:
Overall Officials: Ketty Peris, Prof, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stingeni L, Marietti R, Bianchi L, Guarneri F, Ferrucci SM, Faraci AG, Foti C, Romita P, Patruno C, Napolitano M, Gallo R, Corazza M, Schena D, Milanesi N, Bruni F, Pigatto P, Musumeci ML, Martina E, Piras V, Tramontana M, Hansel K. Patch testing of budesonide in Italy: The SIDAPA baseline series experience, 2018-2019. Contact Dermatitis. 2021 Sep;85(3):317-323. doi: 10.1111/cod.13873. Epub 2021 May 24. PMID 33931866
- [Background] Solberg JBK, Quaade AS, Jacobsen SB, Andersen JD, Kampmann ML, Morling N, Litman T, Thyssen JP, Johansen JD. The transcriptome of hand eczema assessed by tape stripping. Contact Dermatitis. 2022 Feb;86(2):71-79. doi: 10.1111/cod.14015. Epub 2021 Dec 8. PMID 34812515
- [Background] Nakashima C, Yanagihara S, Otsuka A. Innovation in the treatment of atopic dermatitis: Emerging topical and oral Janus kinase inhibitors. Allergol Int. 2022 Jan;71(1):40-46. doi: 10.1016/j.alit.2021.10.004. Epub 2021 Nov 21. PMID 34815171
- [Background] Diepgen TL, Andersen KE, Chosidow O, Coenraads PJ, Elsner P, English J, Fartasch M, Gimenez-Arnau A, Nixon R, Sasseville D, Agner T. Guidelines for diagnosis, prevention and treatment of hand eczema--short version. J Dtsch Dermatol Ges. 2015 Jan;13(1):77-85. doi: 10.1111/ddg.12510. English, German. PMID 25640512
- [Background] Thyssen JP, Schuttelaar MLA, Alfonso JH, Andersen KE, Angelova-Fischer I, Arents BWM, Bauer A, Brans R, Cannavo A, Christoffers WA, Crepy MN, Elsner P, Fartasch M, Filon FL, Gimenez-Arnau AM, Goncalo M, Guzman-Perera MG, Hamann CR, Hoetzenecker W, Johansen JD, John SM, Kunkeler ACM, Hadzavdic SL, Molin S, Nixon R, Oosterhaven JAF, Rustemeyer T, Serra-Baldrich E, Shah M, Simon D, Skudlik C, Spiewak R, Valiukeviciene S, Voorberg AN, Weisshaar E, Agner T. Guidelines for diagnosis, prevention, and treatment of hand eczema. Contact Dermatitis. 2022 May;86(5):357-378. doi: 10.1111/cod.14035. Epub 2022 Mar 3. PMID 34971008
- [Background] Quaade AS, Simonsen AB, Halling AS, Thyssen JP, Johansen JD. Prevalence, incidence, and severity of hand eczema in the general population - A systematic review and meta-analysis. Contact Dermatitis. 2021 Jun;84(6):361-374. doi: 10.1111/cod.13804. Epub 2021 Feb 23. PMID 33548072